CLINICAL TRIAL: NCT04998162
Title: SVF in Infiltrative Therapy for Ankle Osteoarthritis: A Pilot Study
Brief Title: Injections of SVF in Ankle Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADSCs-INT
Record Dates: First submitted 2021-05-18; First posted 2021-08-10 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Ankle Osteoarthritis
Keywords: SVF; ankle; ankle osteoarthritis; stromal vascular fraction; injection treatment; ADSCs; Pilot study; Adipose Derived Stromal Cell's

STUDY DESIGN:
Intervention Model Description: 30 patients with moderate to severe ankle osteoarthritis (Giannini grade 1-3) will be included in the study and the affected ankle will be treated with a single injection of SVF (Stromal vascular fraction). Each patient will sign an informed consent for the participation in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SVF injection (Experimental): All patients with ankle osteoarthritis will be treated with a single injection of SVF, obtained from the patient's abdominal adipose tissue. All patients will be examined with a baseline clinical visit and will be followed-up with clinical evaluation at 1, 3, 6, 12 and 24 months.
  Interventions: Procedure: SVF injection

INTERVENTIONS:
Procedure: SVF injection — Patients with ankle osteoarthritis will be treated with a single injection of 5 cc of SVF (stromal vascular fraction), obtained from patient's abdominal adipose tissue and concentrated through OPTYFAT device. Infiltration of the ankle, occurs from the safest portal, that is, from the antero- medial, between the tibialis anterior and the saphenous vein and nerve at the level of the articular rima.

SUMMARY:
The aim of this pilot study is to analyze the effect of SVF injection produced by adipose tissue processing, in terms of clinical improvement, in patients with moderate to severe (stage 1-3) ankle osteoarthritis. Evaluation will be performed by administering pre-operative and post-operative clinical assessment questionnaires.

Patients will be followed-up with a pre-operative evaluation and post-operative evaluations at 30 days, 3-6-12, and 24 months after application.

DETAILED DESCRIPTION:
30 patients with moderate to severe ankle osteoarthritis (grade 1-3 according to Giannini's classification) will be included in this pilot study, in which patients will be treated with single injection of Stromal Vascular Fraction - SVF ,obtained by processing the patient's abdominal adipose tissue. All patients will be examined with a baseline clinical visit. For obtaining SVF, will be carried out a routinely performed procedure aimed at obtaining a small amount of adipose tissue from all patients. Subsequently, patients will be followed up with clinical evaluation at 1, 3, 6, 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients suffering from moderate to severe unilateral ankle arthrosis (grade 1-3 according to Giannini's classification);
2. Patients who gave written informed consent to participate in the study;
3. .Patients with MRI examination showing absence of osteochondral lesion;
4. Patients who have given their willingness to come to the Institute for follow-up visits

Exclusion Criteria:

1. Patients with BMI>30 kg/m2
2. Patients with Rheumatoid Arthritis
3. Patients with chronic inflammatory joint disease;
4. Patients with acute or chronic infections;
5. Patients with pre-existing abnormalities of gait kinematics (amputations, neuro-muscular diseases, poliomyelitis, hip dysplasia);
6. Patients with severe knee arthrosis (Kellgren-Lawrence>3);
7. Patients with ankle deformities greater than 8°;
8. Patients with pain on other joints of the foot;
9. Patients with severe postural instability;
10. Patients with cognitive deficits;
11. Patients with concomitant neurological pathologies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
AOS (Ankle Osteoarthritis Scale) | Baseline to 24 months
  AOS is a score divided into 2 subscales, each with 9 questions. The first section assesses pain, while the other assesses ankle function. The answers consist of a rating on a 100-mm-long horizontal visual analog scale (from "no pain" to "worst pain imaginable" for pain section, and "no limitation" and "extremely limited" for function section). The highest possible value of the score is 100 (worst score) and the lowest (best score) is 0.

SECONDARY OUTCOMES:
AOFAS (The American Orthopedic Foot and Ankle Score): | baseline, 1,3,6,12,24 months
  AOFAS is the most validated and widely used clinical and functional assessment tool for the ankle and foot. The score consists of 9 questions grouped into 3 categories for a total of 100 points maximum: Pain (up to 40 points), Function (up to 50 points) and Alignment (up to 10 points).100 points represent the best possible clinical-functional condition and absence of symptoms, 0 points represent the worst possible clinical-functional condition. AOFAS is a tool that combines the subjective component of the patients with the objective evaluation by the physician.
VAS-pain (Visual Analogue Scale) | baseline, 1,3,6,12,24 months
  VAS Iis represented by a line 10 cm long: one end indicates the absence of pain and corresponds to 0, the other end indicates the worst pain imaginable and corresponds to 10. The scale is filled by the patient who is asked to draw a mark on the line representing the perceived pain. The distance measured from the 0 end corresponds to the subjective measure of pain
Range Of Motion (ROM) | baseline, 1,3,6,12,24 months
  Baseline and follow-up measurement of ROM range of motion of the treated ankle
SF-12 (12-Item Short Form Survey): | baseline, 1,3,6,12,24 months
  SF-12 consist of 12 questions that permit to investigate the two synthetic indices, PCS Physical Component Summary for the Physical State and MCS Mental Component Summary for the Mental State. The main strengths of this questionnaire are its brevity and relative ease of use.
EQ-5D (EuroQoL) Current Health Assessment | baseline, 1,3,6,12,24 months
  The EQ-5D profile, asks patients to classify their health based on self-assessed levels of problems ("no", "some", "extreme") on five dimensions.
EQ-VAS | baseline, 1,3,6,12,24 months
  EQ-VAS Is a visual analog scale that has a range of scores from 0 (worst imaginable health condition) to 100 (best imaginable health condition).
Patient Acceptable Symptom State (PASS): | baseline, 1,3,6,12,24 months
  A tool to assess patient satisfaction in consideration of their current degree of pain, function, and daily activity. Patients can express if their state of health will be satisfying, answering "yes" or "no.
Final treatment opinion | baseline, 1,3,6,12,24 months
  The patient should indicate satisfaction and relative degree with treatment at the end of the clinical trial (24 months follow-up). All patients will be able to indicate their health condition by choosing from this answers; "Full recovery", "much better", "somewhat better", "no change", "a little worse", "much worse".

CONTACTS AND LOCATIONS:
Overall Officials: Massimiliano Mosca, MD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barfod KW, Blond L. Treatment of osteoarthritis with autologous and microfragmented adipose tissue. Dan Med J. 2019 Oct;66(10):A5565. PMID 31571571
- [Background] Jones IA, Wilson M, Togashi R, Han B, Mircheff AK, Thomas Vangsness C Jr. A randomized, controlled study to evaluate the efficacy of intra-articular, autologous adipose tissue injections for the treatment of mild-to-moderate knee osteoarthritis compared to hyaluronic acid: a study protocol. BMC Musculoskelet Disord. 2018 Oct 24;19(1):383. doi: 10.1186/s12891-018-2300-7. PMID 30355323
- [Background] Shimozono Y, Dankert JF, Kennedy JG. Arthroscopic Debridement and Autologous Micronized Adipose Tissue Injection in the Treatment of Advanced-Stage Posttraumatic Osteoarthritis of the Ankle. Cartilage. 2021 Dec;13(1_suppl):1337S-1343S. doi: 10.1177/1947603520946364. Epub 2020 Aug 6. PMID 32757620
- [Background] Freitag J, Wickham J, Shah K, Tenen A. Effect of autologous adipose-derived mesenchymal stem cell therapy in the treatment of an osteochondral lesion of the ankle. BMJ Case Rep. 2020 Jul 8;13(7):e234595. doi: 10.1136/bcr-2020-234595. PMID 32641315
- [Background] McIntyre JA, Jones IA, Han B, Vangsness CT Jr. Intra-articular Mesenchymal Stem Cell Therapy for the Human Joint: A Systematic Review. Am J Sports Med. 2018 Dec;46(14):3550-3563. doi: 10.1177/0363546517735844. Epub 2017 Nov 3. PMID 29099618
- [Background] Giannini S, Buda R, Faldini C, Vannini F, Romagnoli M, Grandi G, Bevoni R. The treatment of severe posttraumatic arthritis of the ankle joint. J Bone Joint Surg Am. 2007 Oct;89 Suppl 3:15-28. doi: 10.2106/JBJS.G.00544. No abstract available. PMID 17908868